CLINICAL TRIAL: NCT02369159
Title: A Phase 3, Randomized, Open Label, Active-controlled Study to Evaluate the Safety, Pharmacokinetics and Effectiveness of IV Peramivir Compared to Oral Oseltamivir in Pediatric Subjects With Acute Uncomplicated Influenza
Brief Title: Safety, PK and Effectiveness of IV Peramivir Versus Oseltamivir in Pediatric Subjects With Uncomplicated Influenza
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCX1812-305
Record Dates: First submitted 2015-02-17; First posted 2015-02-23 (Estimated); Results first posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-02

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — peramivir; Oseltamivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peramivir (IV) (Experimental): Subjects randomized to peramivir will receive an age appropriate single dose, diluted to a maximum volume of 100 mL in normal saline, administered as a short intravenous infusion over a minimum of 15 minutes.
  * Subjects ≥12 years will receive a dose of 600 mg.
  * Subjects <12 years will receive a dose of 12 mg/kg (to a maximum dose of 600 mg).
  * Subjects < 6 months will receive a dose of 8 mg/kg.
  Interventions: Drug: Peramivir
- Oseltamivir (Active Comparator): Subjects randomized to oral oseltamivir will receive an age appropriate dose twice daily for 5 days.
  * Subjects ≥ 13 years will receive a 75mg dose administered as a capsule or oral suspension (twice daily for 5 days).
  * Subjects < 13 years of age will receive a weight-based dose administered as a capsule or oral suspension (twice daily for 5 days).
  Interventions: Drug: Oseltamivir

INTERVENTIONS:
Drug: Peramivir
  Arms: Peramivir (IV)
Drug: Oseltamivir
  Arms: Oseltamivir

SUMMARY:
This study will evaluate the safety, pharmacokinetics and effectiveness of a single dose of IV peramivir compared to a standard 5 day course of oral oseltamivir in the treatment of pediatric subjects with acute uncomplicated influenza.

ELIGIBILITY:
Key Inclusion Criteria:

1. Clinical signs and symptoms consistent with acute influenza infection consisting of an oral temperature ≥ 100°F (37.8°C) or rectal temperature ≥ 101.3ºF (≥ 38.5ºC) with at least one respiratory symptom (cough or rhinitis) OR Positive influenza determined by PCR or Rapid Antigen Test
2. Onset of symptoms no more than 72 hours before presentation for screening for subjects < 2 years old.

Key Exclusion Criteria:

1. Pregnant or breast-feeding females
2. Development of symptoms while hospitalized
3. Presence of a chronic disease or illness that may indicate increased risk for influenza-related complications
4. Presence of immunocompromised status

Ages: 0 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 137 (Actual)
Dates: Start 2015-03-11 (Actual); Primary Completion 2019-10-28 (Actual); Study Completion 2020-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Vanchiere, MD, PhD, Principal Investigator — Chief, Pediatric Infectious Diseases, Louisiana State University
Locations (10):
- United States (9):
  - Peramivir Investigative Site, Shreveport, Louisiana
  - Peramivir investigative site, Dayton, Ohio
  - Peramivir investigative site, Smithfield, Pennsylvania
  - Peramivir Investigative Site, Houston, Texas
  - Peramivir investigative site, San Antonio, Texas
  - Peramivir investigative site, Splendora, Texas
  - Peramivir investigative site, Draper, Utah
  - Peramivir investigative site, Salt Lake City, Utah
  - Peramivir investigative site, South Jordan, Utah
- Peramivir Investigative Site, Pretoria, South Africa

RESULTS

PARTICIPANT FLOW:
Groups:
- Peramivir: Age-appropriate dose Peramivir, administered as a single short iv infusion:
  Subjects ≥12 years - 600 mg. Subjects <12 years - 12 mg/kg (max. 600 mg). Subjects < 6 months - 8 mg/kg.
- Oseltamivir: Age appropriate oral dose of Oseltamivir BID for 5 days:
  Subjects ≥ 13 years - 75mg dose as a capsule or oral suspension. Subjects < 13 years - weight-based dose as a capsule or oral suspension.
Period: Overall Study
Arm/Group | Peramivir | Oseltamivir
Started | 114 | 23
ITT Population (Intend-to-treat (ITT) population included all randomized subjects) | 114 | 23
Safety Population (Safety Population included all randomized subjects who received ≥ 1 partial dose of peramivir or oseltamivir.) | 107 | 23
ITTI Population (Intent-to-treat-infected (ITTI) population included all subjects who were enrolled, treated, and had influenza confirmed by RT-PCR.) | 81 | 16
E-R Population (Exposure-response (E-R) Population included all subjects in the ITTI population who had a quantifiable peramivir concentration on Day 1 and had ≥ 1 post-baseline effectiveness assessment.) | 80 | 0 (Milestone only applied to Peramivir group)
Completed | 106 | 21
Not Completed | 8 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 7 | 0

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITTI) population included all randomized subjects and was the primary population for analyses of demography and subject accountability.
Groups:
- Peramivir: Age-appropriate single dose Peramivir, administered as a single short iv infusion:
  Subjects ≥12 years - 600 mg. Subjects <12 years - 12 mg/kg (max. 600 mg). Subjects < 6 months - 8 mg/kg.
- Total: Total of all reporting groups
Arm/Group | Peramivir | Oseltamivir | Total
Number analyzed (Participants) | 114 | 23 | 137
Age, Continuous [Mean (Standard Deviation); unit: Age at time of randomisation - years] — Population: Mean age (SD) is reported for the overall ITT population and for each of the 4 age groups
  Age at time of randomisation - years
    Overall | 8.0 (5.07) | 9.9 (4.99) | 8.4 (5.09)
    ≥ 28 days to < 2-year-old cohort: number analyzed (Participants) | 20 | 1 | 21
    ≥ 28 days to < 2-year-old cohort | 1.3 (0.47) | 1.0 (NA) — Only 1 participant in group | 1.3 (0.47)
    ≥ 2 to < 7-year-old cohort: number analyzed (Participants) | 32 | 6 | 38
    ≥ 2 to < 7-year-old cohort | 4.9 (1.47) | 4.7 (1.60) | 4.8 (1.47)
    ≥ 7 to < 13-year-old cohort: number analyzed (Participants) | 39 | 9 | 48
    ≥ 7 to < 13-year-old cohort | 9.6 (1.75) | 9.7 (1.92) | 9.6 (1.76)
    ≥ 13 to < 18-year-old cohort: number analyzed (Participants) | 23 | 7 | 30
    ≥ 13 to < 18-year-old cohort | 15.7 (1.45) | 15.9 (1.50) | 15.7 (1.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 14 | 73
  Male | 55 | 9 | 64
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 0 | 8
  White | 98 | 23 | 121
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 0 | 7
Baseline Influenza Viral Titer [Count of Participants; unit: Participants]
  Positive | 70 | 14 | 84
  Negative | 37 | 9 | 46
  Missing | 7 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability, as Measured by the Number of Participants Experiencing Adverse Events.
Description: Safety evaluation included assessment of Adverse Events (AEs).
Time Frame: 14 days
Population: The Safety population included all randomized subjects who received ≥ 1 partial dose of peramivir or oseltamivir.
Measure: Count of Participants; unit: Participants
Arm/Group | Peramivir | Oseltamivir
Number analyzed (Participants) | 107 | 23
Participants
  Adverse Event | 22 | 5
  Severe or life-threatening Adverse Event | 2 | 0
  Adverse Event possibly, probably, or definitely related to study drug | 8 | 4
  Serious Adverse Events | 0 | 0
  Adverse Event leading to discontinuation from study | 0 | 1
  Adverse Event leading to Death | 0 | 0

2. Secondary Outcome: Plasma Exposure of IV Peramivir as Measured by the Drug Concentration Over 6 Hours Post-dose
Description: Up to 4 blood samples will be drawn, where possible: immediately following infusion and 30 to 60 mins, 1 to 3 hrs and 4 to 6 hrs post-infusions. AUC calculations were performed in Phoenix WinNonlin using the linear/log trapezoidal rule. AUC0-last was calculated between start of the infusion and the time of the last measurable concentration.
Time Frame: up to 6 hours post peramivir infusion
Population: The Intent-to-Treat (ITTI) population included all randomized subjects. Of these 114 subjects, 106 had sufficient PK samples collected for inclusion in the peramivir PK analysis
Measure: Mean (Standard Deviation); unit: ng*h/mL
Groups:
- Peramivir (≥ 28 Days - < 2 Years): Age-appropriate dose Peramivir, administered as a single short iv infusion:
  Subjects <2 years - 12 mg/kg (max. 600 mg). Subjects < 6 months - 8 mg/kg.
- Peramivir (≥ 2 - < 7 Years): 12 mg/kg (max. 600 mg) dose Peramivir, administered as a single short iv infusion
- Peramivir (≥ 7 - < 13 Years): Age-appropriate dose Peramivir, administered as a single short iv infusion:
  Subjects ≥12 years - 600 mg. Subjects <12 years - 12 mg/kg (max. 600 mg).
- Peramivir (≥ 13 - < 18 Years): 600 mg dose Peramivir, administered as a single short iv infusion
Arm/Group | Peramivir (≥ 28 Days - < 2 Years) | Peramivir (≥ 2 - < 7 Years) | Peramivir (≥ 7 - < 13 Years) | Peramivir (≥ 13 - < 18 Years)
Number analyzed (Participants) | 18 | 29 | 39 | 20
ng*h/mL
  AUC0-last | 56200 (21430) | 71200 (31380) | 87000 (40750) | 72400 (19970)
  AUC0-3: number analyzed (Participants) | 15 | 28 | 39 | 20
  AUC0-3 | 53300 (19100) | 68100 (27060) | 81400 (35090) | 68300 (19190)

3. Secondary Outcome: Time to Resolution of Fever
Description: Time for fever resolution based on subject diary record of temperature recorded twice daily. A subject had resolution of fever if he/she had oral temperature of < 99.4°F or an axillary temperature of < 98.4°F and no antipyretic medications were taken for ≥ 12 hours. The time to resolution of fever was estimated for each age group and overall using the Kaplan-Meier method with temperature and symptom relief medication information obtained from the Subject Diary data.
Time Frame: 14 days
Population: Intent to treat infected (ITTI) population. Subjects who did not have resolution of fever were censored at the time of their last non-missing post-baseline temperature assessment; this included 1 subject in the '≥ 28 days - < 2 years' cohort treated with Peramivir. Seventeen subjects were excluded from summaries due to missing data or events resolving prior to initiation of study drug.
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Oseltamivir (≥ 28 Days - < 2 Years); Oseltamivir (≥ 2 - < 7 Years); Oseltamivir (≥ 7 - < 13 Years): Weight-based dose of Oseltamivir as a capsule or oral suspension BID for 5 days.
- Oseltamivir (≥ 13 - < 18 Years): 75mg dose of Oseltamivir as a capsule or oral suspension BID for 5 days.
Arm/Group | Peramivir (≥ 28 Days - < 2 Years) | Oseltamivir (≥ 28 Days - < 2 Years) | Peramivir (≥ 2 - < 7 Years) | Oseltamivir (≥ 2 - < 7 Years) | Peramivir (≥ 7 - < 13 Years) | Oseltamivir (≥ 7 - < 13 Years) | Peramivir (≥ 13 - < 18 Years) | Oseltamivir (≥ 13 - < 18 Years)
Number analyzed (Participants) | 10 | 1 | 21 | 2 | 27 | 5 | 9 | 5
hours | 39.7 (6.55) | 61.8 (NA) — Only one participant in group | 58.8 (8.42) | 16.0 (2.38) | 36.3 (5.00) | 29.7 (7.82) | 51.3 (11.59) | 43.9 (13.67)

4. Secondary Outcome: Time to Resolution of Influenza Symptoms
Description: Subjects or parents or caregivers were asked to provide an assessment of age-appropriate influenza symptoms on a 4-point severity scale (0,absent; 1, mild; 2, moderate; 3, severe) twice daily beginning before screening on Day 1 until symptoms resolved or until the last follow-up visit. Time to alleviation of symptoms was the number of hours from initiation of study drug until the start of the time period in which all age-appropriate symptoms of influenza were either absent or present at a level no greater than mild for at least 21.5 (24 - 10%) hours. Subjects who did not experience alleviation of symptoms were censored at the last observed symptom assessment.
Time Frame: 14 days
Population: Intent to treat infected (ITTI) population. Subjects with no alleviation of symptoms were censored at date of last post-baseline assessment; including 1 subject in the '≥ 28 days to < 2 yrs, Peramivir' group, 1 subject in the '≥ 2 to < 7 yrs, Peramivir' group, 4 subjects in the '≥ 7 to < 13 yrs, Peramivir' group and 1 subject each in the '≥ 13 to < 18 yrs' Peramivir and Oseltamivir groups. Seven subjects were excluded due to missing data or events resolving prior to initiation of study drug.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Peramivir (≥ 28 Days - < 2 Years) | Oseltamivir (≥ 28 Days - < 2 Years) | Peramivir (≥ 2 - < 7 Years) | Oseltamivir (≥ 2 - < 7 Years) | Peramivir (≥ 7 - < 13 Years) | Oseltamivir (≥ 7 - < 13 Years) | Peramivir (≥ 13 - < 18 Years) | Oseltamivir (≥ 13 - < 18 Years)
Number analyzed (Participants) | 10 | 1 | 24 | 2 | 28 | 7 | 13 | 5
hours | 76.1 (19.77) | 98.9 (NA) — Only one participant in group | 94.1 (11.53) | 20.7 (2.32) | 66.6 (7.83) | 134.4 (15.74) | 101.3 (18.46) | 75.5 (12.76)

5. Secondary Outcome: Time to Reduction in Viral Shedding
Description: Assessment of viral shedding in bilateral, mid-nasal swab specimens taken at baseline and then on Day 3, 7 and 14.
Time Frame: 14 days
Population: Intent to treat infected (ITTI) population + ITT population with positive baseline influenza viral titers [> 0.5 log10 TCID50/mL]; a total of 84 subjects.
Measure: Number; unit: participants with positive viral titer
Arm/Group | Peramivir (≥ 28 Days - < 2 Years) | Oseltamivir (≥ 28 Days - < 2 Years) | Peramivir (≥ 2 - < 7 Years) | Oseltamivir (≥ 2 - < 7 Years) | Peramivir (≥ 7 - < 13 Years) | Oseltamivir (≥ 7 - < 13 Years) | Peramivir (≥ 13 - < 18 Years) | Oseltamivir (≥ 13 - < 18 Years)
Number analyzed (Participants) | 8 | 1 | 23 | 2 | 27 | 6 | 12 | 5
participants with positive viral titer
  Baseline | 8 | 1 | 23 | 2 | 27 | 6 | 12 | 5
  Day 3: number analyzed (Participants) | 8 | 1 | 22 | 1 | 27 | 6 | 12 | 5
  Day 3 | 6 | 1 | 12 | 1 | 13 | 6 | 6 | 2
  Day 7: number analyzed (Participants) | 8 | 1 | 23 | 1 | 26 | 6 | 12 | 5
  Day 7 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0
  Day 14: number analyzed (Participants) | 8 | 1 | 23 | 1 | 26 | 6 | 12 | 5
  Day 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Changes in Influenza Virus Titer in Nasopharyngeal Samples in Response to Treatment.
Description: Change in influenza viral titers was defined as the time-weighted change from Baseline in log_10 tissue culture infective dose_50 (TCID50/mL) and was summarized for each treatment group.
Time Frame: Change from baseline assessed on days 3, 7 and 14.
Population: The Intent To Treat Infected (ITTI) population included all subjects who were enrolled, received study drug, and had confirmed influenza A and/or B by PCR. Thirteen subjects were excluded due to a negative or missing baseline titer.
Measure: Median (Full Range); unit: influenza viral titer - log10 TCID50/mL
Arm/Group | Peramivir | Oseltamivir
Number analyzed (Participants) | 70 | 14
influenza viral titer - log10 TCID50/mL
  Baseline | 4.38 [0.75 to 6.50] | 4.50 [1.50 to 5.75]
  Day 3 - Change rom baseline | -2.75 [-6.00 to 2.50] | -3.25 [-5.00 to 1.25]
  Day 7 - Change from baseline | -3.75 [-6.00 to 1.00] | -4.00 [-5.25 to -1.00]
  Day 14 - Change from baseline | -3.75 [-6.00 to -0.25] | -4.00 [-5.25 to -1.00]

7. Secondary Outcome: Influenza-Related Complications Assessment.
Description: The investigator performed a full physical exam at baseline. At each follow-up visit, study personnel evaluated the subject for the presence of clinical signs and symptoms of the following influenza-related complications: sinusitis, otitis media, bronchitis, and pneumonia requiring antibiotic use, diagnosed after initiation of treatment.
Time Frame: 14 days
Population: Intent-to-treat infected (ITTI) population
Measure: Count of Participants; unit: Participants
Arm/Group | Peramivir | Oseltamivir
Number analyzed (Participants) | 81 | 16
Participants
  Otitis | 3 | 0
  Sinusitis | 2 | 0
  Bronchitis | 0 | 0
  Pneumonia | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs were recorded on Day 1, Day 3, Day 7 and Day 14/Early Withdraw visit.
Description: Adverse events were graded through use of the Division of Acquired Immune Deficiency Syndrome (DAIDS) Tables for Grading Adult and Pediatric Adverse Experiences. Influenza-related complications were not considered AEs unless they met the criteria for an SAE.
Arm/Group | Peramivir | Oseltamivir
All-Cause Mortality (participants affected / at risk) | 0/107 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/107 | 0/23
Other Adverse Events (participants affected / at risk) | 22/107 | 5/23
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peramivir (N=107) | Oseltamivir (N=23)
Vomiting (Gastrointestinal disorders) | 4 (4) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Tympanic membrane hyperaemia (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Elevated aspartate aminotransferase (Investigations) | 2 (2) | 0 (0)
Elevated blood lactate dehydrogenase (Investigations) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Injection site coldness (General disorders) | 1 (1) | 0 (0)
Injection site paraesthesia (General disorders) | 1 (1) | 0 (0)
Injection site rash (General disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tympanic membrane disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Carbon dioxide decreased (Investigations) | 1 (1) | 0 (0)
Psychomotor hyperactivity (Nervous system disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-11-05): https://cdn.clinicaltrials.gov/large-docs/59/NCT02369159/Prot_000.pdf
  • Statistical Analysis Plan (2016-07-11): https://cdn.clinicaltrials.gov/large-docs/59/NCT02369159/SAP_001.pdf